CLINICAL TRIAL: NCT01258556
Title: The Impact of Probiotic Bacteria on the Efficacy of Anti-retroviral Therapy and Recurrence of Bacterial Vaginosis
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Gregor Reid, Lawson Health Research Institute
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 919
Record Dates: First submitted 2010-12-10; First posted 2010-12-13 (Estimated); Last update posted 2010-12-13 (Estimated); Status verified 2010-12

CONDITIONS: Bacterial Vaginosis
MeSH Terms: conditions — Vaginosis, Bacterial

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Probiotic yogurt (Experimental)
  Interventions: Dietary Supplement: Yogurt supplemented with L. rhamnosus fiti
- Placebo yogurt. (Placebo Comparator)
  Interventions: Dietary Supplement: Yogurt not supplemented with a probiotic strain.

INTERVENTIONS:
Dietary Supplement: Yogurt supplemented with L. rhamnosus fiti — 200 ml of L. rhamnosus fiti at 10*9 cfu/ml daily for 30 days.
  Arms: Probiotic yogurt
Dietary Supplement: Yogurt not supplemented with a probiotic strain. — 200 ml yoghurt without L. rhamnosus fiti daily for 30 days.
  Arms: Placebo yogurt.

SUMMARY:
Purpose of the proposed research is to determine the impact of probiotic yogurt supplemented with Lactobacillus rhamnosus (Fiti) compared to regular yogurt on the well-being of women living with HIV.

ELIGIBILITY:
Inclusion criteria:

* Confirmed HIV infection;
* Being treated with anti-retroviral medication for > 6 months.

Exclusion criteria:

* Pregnancy;
* Hypersensitive to fermented milk;
* Intolerant for lactose;
* Complaints of bacterial vaginosis requiring treatment

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2010-06; Primary Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Vaginal microbiota of HIV patients. | 30 days

SECONDARY OUTCOMES:
Bacterial vaginosis. | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Nicodemus Butamanya, MD, Principal Investigator — Sekou-Toure Regional Hospital
Locations (1):
- Sekou-Toure Regional Hospital, Mwanza, Tanzania